CLINICAL TRIAL: NCT00713258
Title: A 24-week, International, Multi Centre, Randomised, Double-blind, Double-dummy, Parallel Group, Phase IV Clinical Trial Investigating Changes in Back Pain in Postmenopausal Women With an Osteoporosis Related Vertebral Fracture(s) Treated With Either 100 µg PTH(1-84) Daily or 70 mg Alendronate Weekly
Brief Title: The Effect of PTH(1-84) or Alendronate on Reduction of Back Pain in Postmenopausal Women With an Osteoporosis Related Vertebral Fracture(s) (FP-005-IM)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrolment
Sponsor: Nycomed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FP-005-IM
Record Dates: First submitted 2008-07-02; First posted 2008-07-11 (Estimated); Results first posted 2011-10-07 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Back Pain
Keywords: Postmenopausal women; Back pain; Osteoporosis related fracture
MeSH Terms: conditions — Back Pain | interventions — Parathyroid Hormone; Alendronate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PTH (1-84) (Active Comparator): PTH (1-84) + placebo alendronate
  Interventions: Drug: Parathyroid hormone (PTH) (1-84)
- Alendronate (Active Comparator): PTH (1-84) placebo + alendronate
  Interventions: Drug: Alendronate

INTERVENTIONS:
Drug: Parathyroid hormone (PTH) (1-84) — 100 µg PTH(1-84) daily
  Arms: PTH (1-84)
Drug: Alendronate — 70 mg alendronate weekly
  Arms: Alendronate

SUMMARY:
The primary objective of this trial is to show that PTH(1-84) is superior to alendronate in reducing back pain intensity over a 24-week treatment period in postmenopausal women with an osteoporosis related vertebral fracture(s).

Secondly the objectives are to investigate any differences in patient reported outcomes between the two treatment arms over a 24-week treatment period in postmenopausal women with an osteoporosis related vertebral fracture(s).

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with a T-score ≤ -1.5 SD and at least one osteoporosis related vertebral fracture. Chronic back pain.

Exclusion Criteria:

* Previous/current treatment and medical history.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2008-04; Primary Completion 2010-05 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nycomed, Roskilde, Denmark

RESULTS

PARTICIPANT FLOW:
Groups:
- PTH (1-84): PTH (1-84) + placebo alendronate
  * PTH (1-84): powder and solvent for solution for injection
  * placebo alendronate: capsule
- Alendronate: PTH (1-84) placebo + alendronate
  * PTH (1-84) placebo: powder and solvent for solution for injection
  * alendronate: capsule
Period: Overall Study
Arm/Group | PTH (1-84) | Alendronate
Started | 41 | 34
Completed | 36 | 28
Not Completed | 5 | 6
Not completed — Adverse Event | 2 | 4
Not completed — Non-Compliance | 2 | 1
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PTH (1-84) | Alendronate | Total
Number analyzed (Participants) | 41 | 34 | 75
Age Continuous [Mean (Standard Deviation); unit: years] | 70.7 (9.14) | 69.8 (7.84) | 70.3 (8.53)
Sex/Gender, Customized [Number; unit: participants]
  Female | 41 | 34 | 75
Vertebral Fracture at Baseline [Mean (Standard Deviation); unit: vertebral fractures per patient] — The baseline measure is shown as average number per patient.
  vertebral fractures per patient | 3.44 (2.49) | 2.94 (1.97) | 3.21 (2.27)
Family history of osteoporosis [Number; unit: patients] — A family history of osteoporosis was reported by 22 subjects, which differs from the overall number of baseline participants.
  patients | 13 | 9 | 22
Age at onset of menopause [Mean (Standard Deviation); unit: years] | 48.5 (3.68) | 48.6 (5.25) | 48.5 (4.43)
Mean NRS score [Mean (Standard Deviation); unit: scores on a scale] — NRS = 11-point numerical rating scale to assess the pain. The NRS score ranges from 0 to 10, with lower scores meaning less pain.
  scores on a scale | 6.60 (1.45) | 6.36 (1.70) | 6.49 (1.56)

OUTCOME MEASURES:

1. Primary Outcome: Change in Back Pain Intensity During 24 Weeks of Treatment Using a Numerical Rating Scale.
Description: The daily patient assessment of intensity of back pain is based on the Numerical Rating Scale (NRS) which is an 11-point numerical rating scale (from 0-10 with 0 = "no pain" and 10 = "unendurable pain").
Time Frame: Baseline and 24 weeks treatment
Population: The number of participants analyzed is "0", because the reduction of the sample size from 300 to 75 subjects due to early trial termination resulted in a small number of subjects with data available. This is far below the number needed to demonstrate a significant difference between the comparison groups and the data have no statistical validity.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | PTH (1-84) | Alendronate
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Physical Disability and Patient Reported Outcomes During 24 Weeks of Treatment
Description: Three times during the trial the patients will be asked how their pain affects their ability to manage everyday life. This information will be collected by use of the Oswestry Disability Index (ODI) questionnaire. The questions relate to daily life activities and indicate to what extent a person's functional level is restricted by pain.
  ODI scores from 0 = "no disability" to 100 = "maximum disability".
  Patient reported outcomes will be assessed by using two questionnaires related to health status and quality of life status.
Time Frame: Baseline and 24 weeks treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | PTH (1-84) | Alendronate
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: The safety analysis set was defined as all subjects that were randomized and given at least 1 dose of the Investigational Medicinal Product (IMP). Subjects were analysed as treated. The safety set is equivalent with the Intention-to-treat (ITT) set.
Arm/Group | PTH (1-84) | Alendronate
Serious Adverse Events (participants affected / at risk) | 1/41 | 5/34
Other Adverse Events (participants affected / at risk) | 18/41 | 13/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PTH (1-84) (N=41) | Alendronate (N=34)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PTH (1-84) (N=41) | Alendronate (N=34)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) — non-serious
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 10 (11) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After publication of the results or 24 months after Clinical Trial Report has been finalised, whichever comes first, Nycomed acknowledge the Investigator's rights to publish results from this trial. Any such scientific paper, presentation, communication or other information concerning the trial described in this protocol must be submitted to Nycomed for review prior to submission for publication/presentation. Review comments will be given within a month from receipt of the manuscript.